CLINICAL TRIAL: NCT00226993
Title: Phase I/II Study of Intratumoral Injection of CPG 7909, A TLR9 Agonist, Combined With Local Radiation for Patients With Recurrent Mycosis Fungoides
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ronald Levy, Robert K. and Helen K. Summy Professor in the School of Medicine, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYMNHL0021; 95850; LYMNHL0021; NCT00226993
Record Dates: First submitted 2005-09-13; First posted 2005-09-27 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides | interventions — ProMune

INTERVENTIONS:
Drug: CPG 7909

SUMMARY:
This is a single institution phase I / II trial to evaluate the safety and efficacy of intratumoral CpG injections combined with local radiation in patients with mycosis fungoides. Patients will receive low-dose radiotherapy to a single tumor site on days 1 and 2 (2 Gy each day). CpG injections will be administered into the same tumor site within 24 hours before or 24 hours after each radiation treatment. Weekly doses of (intratumoral or peritumoral injections) CpG will be then administered subcutaneously in the region of previous injections for 23 additional doses. The total treatment duration is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:- Biopsy confirmed mycosis fungoides of stage IB-IVA. Patients must have failed or have been intolerant of at least 2 topical or one systemic treatment.

* Patients must have at least one site of disease that is accessible for intratumoral injection of CpG percutaneously, and the second site to follow treatment response.
* 18 years of age or older
* Karnofsky Performance Status (KPS) of > 70.
* Adequate bone marrow function: WBC>4,000uL, hemoglobin > 10g/dL; platelet count >100,000/mm^3; ANC> 1000.
* Adequate hepatic function: bilirubin <= 1.5 mg/dL; SGOT/SGPT<3xupper limit of normal
* Adequate renal function: serum creatinine <= 2.0mg/dL.
* Required wash out periods for prior therapy:

  * Topical therapy: 2 weeks
  * Chemotherapy: 4 weeks
  * Radiotherapy (including photo therapy): 4 weeks
  * Systemic biological therapy for mycosis fungoides: 4 weeks
  * Other investigational therapy: 4weeks
* Patients of reproductive potential and their partners must agree to use an effective (>90% reliability) form of contraception during the study and for 4 weeks following the last study drug administration.
* Women of reproductive potential must have negative urine pregnancy test.
* Life expectancy greater than 4 months.
* Able to comply with the treatment schedule. Exclusion Criteria:- Pre-existing autoimmune or antibody mediated disease including: systemic lupus, erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, but excluding controlled thyroid disease, or the presence of autoantibodies without clinical autoimmune disease.
* Known history of human immunodeficiency virus (HIV), hepatitis B or hepatitis C (active, prior treatment, or both).
* Patients with active infection or with a fever >38.50 C within three days prior to the first scheduled treatment.
* CNS metastases
* Prior malignancy (active within 5 years of screening) except basal cell or completely excised non-invasive squamous cell carcinoma of the skin, or in situ squamous cell carcinoma of the cervix.
* Prior treatment with CpG.
* History of allergic reactions attributed to compounds of similar composition to CPG 7909
* Current anticoagulant therapy (ASA<= 325mg/day allowed).
* Significant cardiovascular disease (i.e. NYHA class 3 congestive heart failure; myocardial infarction with the past 6 months; unstable angina; coronary angioplasty with the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias).
* Pregnant or lactating.
* Any other medical history, including laboratory results, deemed by the investigator to be likely to interfere with their participation in the study, or to interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-03; Primary Completion 2006-12 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy of intratumoral CpG injections combined with local radiation

SECONDARY OUTCOMES:
To determine local and systemic anti-tumor effect.
To evaluate tumor-specific humoral and cellular immune responses

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Levy, Principal Investigator — Stanford University

REFERENCES:
- [Derived] Kim YH, Gratzinger D, Harrison C, Brody JD, Czerwinski DK, Ai WZ, Morales A, Abdulla F, Xing L, Navi D, Tibshirani RJ, Advani RH, Lingala B, Shah S, Hoppe RT, Levy R. In situ vaccination against mycosis fungoides by intratumoral injection of a TLR9 agonist combined with radiation: a phase 1/2 study. Blood. 2012 Jan 12;119(2):355-63. doi: 10.1182/blood-2011-05-355222. Epub 2011 Nov 1. PMID 22045986